CLINICAL TRIAL: NCT00605124
Title: Progressive Exercise After Total Knee Arthroplasty: A Randomised Controlled Trial
Brief Title: Progressive Exercise After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Mirja Vuorenmaa, physiotherapist, Jyväskylä Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSSHP Dnro6/2007; KSSHP (Other: KSSHP)
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; total knee arthroplasty; exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Experimental): progressive exercise, home-based exercise program, tree exercise sessions weekly, chec-up visits every third month
  Interventions: Other: Knee muscle exercises
- Conventional treatment (Active Comparator): Normal treatment, single guidance to home exercise
  Interventions: Other: Knee muscle exercises

INTERVENTIONS:
Other: Knee muscle exercises — Home exercises three times a week, control every three months

SUMMARY:
Total knee arthroplasty (TKA) is performed more than 7.000 times a year in Finland most often for osteoarthritis (OA). While pain is predictably reduced, function does not typically ever reach that of age-matched, uninjured subjects. Quadriceps weakness has been implicated in the development and progression of knee OA and is a significant problem after TKA. Advance to return to normal daily activities is not sufficient to restore knee function or quadriceps strength after TKA.

The aim of this study is to assess the effectiveness of progressive exercise program restoring knee strength, mobility and improving the functional outcome after primary TKA.

DETAILED DESCRIPTION:
Many studies have shown, that after TKA pain decreased significantly, but muscle strength of the operated knee did not recover and may stay under the preoperative level. To find out the effects of progressive exercise program the investigators will perform, 6 weeks after TKA, a randomized clinical trial of lower extremity strength training using two subgroups of people: traditional exercise group and progressive exercise group.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral TKA for knee osteoarthritis

Exclusion Criteria:

* Rheumatoid arthritis
* Fibromyalgia
* Bilateral TKA
* Heart or lung disease, which prevent training
* Unstable serious disease (cancer)
* Reduced cooperation (drug, alcohol abuse, mental illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Functional tests, pain | baseline , 6 weeks after operation (start of training), after 12 months training
  Timed-Up and Go-test, Visual analogue scale (VAS)

SECONDARY OUTCOMES:
Knee muscle strength | baseline, 6 weeks after operation (start of training), after 12 months training
  isometric strength of quadriceps and hamstrings
Health related quality of life | baseline and 12 months
  SF-36
gait analysis | baseline, 6 weeks postoperatively, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD, PhD, Study Director — Central Finland Health Care District; Arja Häkkinen, PhD, Professor, Study Chair — Central Finland Health Care District; Petri Salo, M.Sc., Principal Investigator — Central Finland Health Care District; Mirja Vuorenmaa, M.Sc., Principal Investigator — Central Finland Health Care District; Maija Pesola, MD, Study Chair — Central Finland Health Care District
Locations (1):
- Ceneral Finland Health Care District, Jyväskylä, Finland